CLINICAL TRIAL: NCT00784524
Title: A Phase II Study of Allogeneic Large Multivalent Immunogen (LMI) Vaccine and IL-2 for the Treatment of Stable Metastatic Breast Cancer
Brief Title: Phase II Study of Allo LMI Vaccine With IL-2 for Stable Metastatic Breast Ca
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007LS094; 0802M25946 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-11-01; First posted 2008-11-04 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LMI Vaccination + IL-2 (Experimental): Patients receiving allogeneic large multivalent immunogen breast cancer vaccine and aldesleukin.
  Interventions: Biological: allogeneic large multivalent immunogen breast cancer vaccine; Biological: aldesleukin

INTERVENTIONS:
Biological: allogeneic large multivalent immunogen breast cancer vaccine — Allogeneic large multivalent immunogen breast cancer vaccine (1 x 10^7, 5-μm silica spheres) will be given as an intradermal injection every 28 days (+/- 3 days). Each vaccine dose will be 0.2 ml.
  Other Names: LMI
Biological: aldesleukin — Subcutaneous aldesleukin (10 x 10^6 International Units) will be given on day 7 and day 8 after each LMI injection.
  Other Names: Interleukin-2; IL-2; Proleukin

SUMMARY:
RATIONALE: Vaccines may help the body build an effective immune response to kill tumor cells. Aldesleukin may stimulate the white blood cells to kill breast cancer cells. Giving vaccine therapy together with aldesleukin may be a more effective treatment for metastatic breast cancer.

PURPOSE: This phase II trial is studying how well giving vaccine therapy together with aldesleukin works in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of allogeneic large multivalent immunogen (LMI) vaccine and aldesleukin, as defined by clinical benefit rate (percentage of patients demonstrating a complete response, partial response, or disease stabilization as assessed by RECIST criteria), in women with stable metastatic breast cancer.

Secondary

* To measure the immune response in patients treated with this regimen.
* To determine the progression-free survival of patients treated with this regimen.
* To determine the 1- and 2-year overall survival rates in patients treated with this regimen.
* To determine the safety profile and toxicity of this regimen in these patients.

OUTLINE: Patients receive allogeneic large multivalent immunogen (LMI) vaccine intradermally on day 1 and aldesleukin subcutaneously on days 7 and 8. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression after 2 courses of vaccine therapy resume the chemotherapy regimen for which prior disease stabilization was achieved. Beginning 2-4 days after completion of chemotherapy, patients receive one dose of LMI vaccine followed by aldesleukin on days 7 and 8. Patients achieving at least stable disease continue to receive LMI vaccine and aldesleukin as above. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Peripheral blood mononuclear cell samples are collected periodically for research studies. Samples are analyzed to assess the frequency of leukocyte subsets (including B cells, T cells, NK cells, and monocytes) via flow cytometry; frequency of T-regs (T cells that express CD4, CD25, and FoxP3); and responses to keyhole limpet hemocyanin and tetanus toxoid via ELISA assay. Other immunological studies are also performed.

After completion of study therapy, patients are followed every 3 months.

ELIGIBILITY:
Inclusion criteria:

* Stage IV, metastatic breast cancer, confirmed by histology or cytology.

  * Disease must be refractory to hormone therapy for tumors that estrogen and/or progesterone receptor positive
  * Disease must be refractory to trastuzumab for tumors that are HER2 positive
  * Disease must be responsive to chemotherapy such that regression or at least stabilization occurs

    * Stable disease is defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease
    * Measurement of regressed or stable disease must be confirmed by repeat evaluation no less than 4 weeks after the initial determination.
* Prior systemic chemotherapy, immunotherapy, biological therapy, or investigational drug therapy is allowed if at least 4 weeks since last treatment.

  * Patient must recover from the acute toxic effects of the treatment prior to study enrollment.
  * There is no limit as to the number of previous chemotherapy regimens received.
* Disease status may be measurable or non-measurable
* Karnofsky performance status >70%
* Women, age 18 years or older
* Adequate organ function within 14 days of study registration including the following:

  * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥ 1.5 x 10^9/L, platelets ≥75 x 10^9/L, and hemoglobin ≥ 8.0 g/dL
  * Hepatic: bilirubin ≤ 3 times the upper limit of normal (× ULN) for patients without tumor involvement of the liver and ≤ 5 X ULN for patients with tumor involvement of the liver; aspartate transaminase (AST) ≤ 2.5 × ULN for patients without tumor involvement of the liver and ≤ 5 X ULN for patients with tumor involvement of the liver
  * Renal: creatinine ≤ 2.0 mg/dL
* Must share at least one class I HLA allele with the HLA-type SKBR3 cell (class I alleles A2, A3, B14, B40, C3, C8)
* Meets eligibility criteria for and agrees to enroll in "MT1999-06: Vaccination with Tetanus Toxoid and Keyhole Limpet Hemocyanin (KLH) to Assess Antigen-Specific Immune Responses" (IRB # 9904M01581, CPRC #2002LS032). Patients who have had tetanus toxoid within the last 7 years will not receive the tetanus vaccine component. For patients who do not know the year of their last tetanus vaccine, tetanus toxoid will be given per protocol. Subjects allergic to seafood will not be co-enrolled into MT1996-06.
* Women of childbearing potential and their partners are required to use an effective method of contraception (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study and for 3 months after the last dose of study drug.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion criteria:

* History of untreated or active brain metastases or positive brain scan at enrollment. Patients with previously treated brain metastases are eligible if stable by CT or MRI for at least 3 months.
* Concurrent malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix
* Active infection
* Solid organ transplantation or autoimmune diseases requiring systemic immunosuppressive therapy; however, topical or inhalational steroids are allowed.
* Symptomatic pulmonary disease (symptoms of dyspnea or rales, wheezes or rhonchi on physical exam) will require pulmonary function testing (PFTs). Those with FEV1 <50% of predicted or corrected DLCO <50% are not eligible.
* Patients with cardiac disease such as recent myocardial infarction (< 3 months prior), unstable angina, or heart failure requiring medical intervention will undergo cardiac evaluation. Cardiac testing may include ECG, MUGA or echocardiogram, and/or thallium stress test as indicated to evaluate cardiac risks. Those patients with exercise-induced ischemia or an ejection fraction by MUGA or echocardiogram < 40% are not eligible.
* Hypersensitivity to any component of the vaccine, including Thimerosal, a mercury derivative, is a contraindication (taken from tetanus toxoid package insert).
* The occurrence of any type of neurologic symptoms to tetanus vaccine in the past is a contraindication to further use (taken from tetanus toxoid package insert).
* Pregnant (positive pregnancy test) or lactating women. Use of LMI vaccine during pregnancy is not approved for use by the FDA during pregnancy. IL-2 is pregnancy category C - risk in pregnancy cannot be ruled out.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Yee, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LMI Vaccination + IL-2
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LMI Vaccination + IL-2
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Response
Description: Percentage of patients achieving complete response, partial response, or disease stabilization as assessed by Response Evaluation Criteria In Solid Tumors Criteria (RECIST) criteria for measurable target lesions and non-measurable non-target lesions assessed by CT, PET-CT or MRI: Complete Response (CR), Disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions or persistence of one or more non-target lesions; Disease Stabilization (SD), Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease; Progressive Disease (PD), >=20% increase in the sum of the longest diameter of target lesions or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | LMI Vaccination + IL-2
Number analyzed (Participants) | 14
Participants | 0

2. Secondary Outcome: Immune Response
Description: Immune responses will be assessed by DTH responses to LMI, IFN-gamma production by CD8+ T cells using the ELISPOT assay, and CD8+ T cell binding to HLA-A2 multimers complexed with breast cancer-derived peptides (multimer analysis).
Time Frame: 48 hours
Population: ELISpot assays were not run because the HLA-multimer assay did not show any strong responses. As such, only DTH responses to LMI were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | LMI Vaccination + IL-2
Number analyzed (Participants) | 13
Participants | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression free survival will be measured in months from time of response to time of disease progression as defined by RECIST (appendix II), "at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s)."
Time Frame: Up to 1 year
Population: One patient's disease had not progressed by the time the study-specified follow-up period had ended and was not included in the analysis..
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | LMI Vaccination + IL-2
Number analyzed (Participants) | 13
months | 4 [3 to 9]

4. Secondary Outcome: Overall Survival
Description: Number of participants alive at one year
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | LMI Vaccination + IL-2
Number analyzed (Participants) | 14
Participants | 11

5. Secondary Outcome: Overall Survival
Description: Number of participants alive at 2 years
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | LMI Vaccination + IL-2
Number analyzed (Participants) | 14
Participants | 8

ADVERSE EVENTS:
Arm/Group | LMI Vaccination + IL-2
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LMI Vaccination + IL-2 (N=14)
Anxiety (Nervous system disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Thrombus/Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LMI Vaccination + IL-2 (N=14)
Elevated Alkaline Phosphatase (Investigations) | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Alanine Aminotransferase Increased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Bronchospasm, Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Chelitis (Skin and subcutaneous tissue disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Fever (General disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dehydration (Gastrointestinal disorders) | 1
Lymphedema (Vascular disorders) | 1
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 3
Candida Intertrigo (Infections and infestations) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Edema: Limb (Vascular disorders) | 4
Jittery (Nervous system disorders) | 1
Fatigue (General disorders) | 9
Flu-Like Syndrome (General disorders) | 7
Flushing (General disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Burping (Gastrointestinal disorders) | 1
Early Satiety (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 7
Heartburn (Gastrointestinal disorders) | 1
Low Hemoglobin (Blood and lymphatic system disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hot Flashes (Vascular disorders) | 2
Pneumonia (Infections and infestations) | 1
Oral Thrush (Infections and infestations) | 1
Chronic Sinusitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3
Infection at Surgery Site (Infections and infestations) | 1
Injection Site Reaction (General disorders) | 8
Insomnia (Psychiatric disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Hyperlipidemia (Investigations) | 1
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Left Foot Drop (Nervous system disorders) | 1
Limited Range of Motion Left shoulder (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Left Foot Cooler than Right (Vascular disorders) | 1
Euphoria (Psychiatric disorders) | 1
Peripheral neuropathy (Nervous system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 1
Vocal Cord Spasm/Dysfunction (Respiratory, thoracic and mediastinal disorders) | 1
Vision Problems, NOS (Eye disorders) | 1
Left Visual Hemianopia (Eye disorders) | 1
Corneal Dystrophy (Eye disorders) | 1
Macular Degeneration (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Bone Pain, NOS (Musculoskeletal and connective tissue disorders) | 2
Chest Pain (General disorders) | 3
Extremity Pain (Musculoskeletal and connective tissue disorders) | 4
Eye Pain (Eye disorders) | 1
Headache (Nervous system disorders) | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 7
Liver Pain (Gastrointestinal disorders) | 1
Muscle Pain (Musculoskeletal and connective tissue disorders) | 3
Oral Cavity Pain (Gastrointestinal disorders) | 1
Pain on Ambulation (Musculoskeletal and connective tissue disorders) | 1
Body Aches (Musculoskeletal and connective tissue disorders) | 3
Heart Palpitations (Cardiac disorders) | 1
Petechiae, Lower Extremity (Skin and subcutaneous tissue disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Erythema, Lower Extremity (Skin and subcutaneous tissue disorders) | 1
Generalized Body Erythema (Skin and subcutaneous tissue disorders) | 1
Chills (General disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 1
Sweating (General disorders) | 1
Taste Alteration (Gastrointestinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Weight Loss (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No